CLINICAL TRIAL: NCT03413358
Title: A Randomized, Controlled, Multicenter Clinical Trial to Evaluate the Efficacy and Safety of Sheng Bai Oral Liquid in Prevention and Treatment for The Decrease of Neutrophils After Chemotherapy in Patients With Non-Small-Cell Lung Cancer
Brief Title: Clinical Trial for Post-marketing Evaluation of Sheng Bai Oral Liquid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BeiJing Yijiayi Medicine Techonoloy Co., Ltd. (Industry)
Collaborators: Hubei Mon Yan Pharmaceutical Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-133-KY-01
Record Dates: First submitted 2018-01-17; First posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Non-small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Cisplatin

STUDY DESIGN:
Intervention Model Description: These subjects will be randomized (1:1) to treatment group or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Platinum-based two medicine (carboplatin / cisplatin) plus Sheng Bai oral liquid.
  Interventions: Drug: Sheng Bai oral liquid; Drug: Platinum-based two medicine (carboplatin / cisplatin) .
- Control group (Experimental): Blank control and Platinum-based two medicine (carboplatin / cisplatin) .
  Interventions: Drug: Platinum-based two medicine (carboplatin / cisplatin) .

INTERVENTIONS:
Drug: Sheng Bai oral liquid — Drug: Sheng Bai oral liquid 40 mL, oral use, thrice daily after screening on the same day in the second course of the chemotherapy.
  Subjects will be treated for 2 courses
  Arms: Treatment group
Drug: Platinum-based two medicine (carboplatin / cisplatin) . — Using Platinum-based two medicine (carboplatin / cisplatin)

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of Sheng Bai oral liquid in prevention and treatment of the decrease of neutrophilics after chemotherapy in patients with non-small-cell lung cancer.

DETAILED DESCRIPTION:
The Clinical trail is a multicenter, prospective, randomized controlled study. The planned sample size is 240 subjects. These subjects will be randomized (1:1) to treatment group (Platinum-based two medicine (carboplatin / cisplatin) plus Sheng Bai oral liquid) or control group ( Platinum-based two medicine (carboplatin / cisplatin) plus blank control). The study population includes the patients with non-small-cell lung cancer .

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are confirmed no small cell lung cancer in accordance with the clinical diagnostic criteria , or by pathological histology or cytology examination which investigators think are suitable to accept The platinum-based doublet chemotherapy（According to RECIST V1.1,patients with no small cell cancers should have one measurable lesions at least ）.
2. ECOG performance status ≤2.
3. Laboratory inspection basically meets the following requirements： 1)Blood test：a. WBC≥ 4.0×109/L, b. ANC≥2.0×109/L, c. PLT≥100×109/L. 2)Biochemical test：a. ALT≤2.5 times the ULN;b. AST≤2.5 times the ULN ;c. Cr<=1.5 times the ULN.
4. Expected survival period is more than 3 months
5. Subjects join the study voluntarily, sign a consent form, have good compliance, and comply with follow-up.

Exclusion Criteria:

1. Patients need radiotherapy, targeted therapy, and other anti-cancer therapies during the trial.
2. Patients accepted radiation in the past 4 weeks before enrollment.
3. Previous bone marrow or stem cell transplant, or organ allograft.
4. Recently severe acute infection is not controlled; purulent or chronic infection is present and the wound is not healed.
5. Patients were or being suspected to be allergic to test drugs or related components.
6. Patients with hypersplenism, hyperthyroidism, adrenal cortical hypofunction, connective tissue disease, infectious diseases, such as viral hepatitis, tuberculosis infection and other diseases which can lead to the decrease of the white blood cells at the same time.
7. Patients with the symptoms of digestive system, such as nausea, vomiting, diarrhea, etc., that are not controlled will influence the test drug.
8. The central nervous system is metastatic and has symptoms.
9. History of another malignancy, except for in situ carcinoma of the cervix, adequately treated basal cell skin carcinoma.
10. Patients with severe heart, liver and kidney diseases; serious diseases of hematopoietic system; bleeding tendency.
11. Patients have a history of drug abuse and cannot be reined ;Patients with symptomatic, uncontrolled nervous disorders, mental illness or psychiatric disorder have less compliance.
12. Female patient is pregnant or breast-feeding, and those patients at childbearing age who are not willing to use methods of contraception.
13. Patients who are currently included in other clinical trials or accepted any experimental drugs in the past 4 weeks.
14. Any condition, in the investigator's opinion, is not in the best interest of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
The incidence and degree of neutropenia after chemotherapy | six weeks
  Comparison of the incidence and extent of neutrophil reduction in two chemotherapy cycles between two groupschemotherapy cycles between two groups according to CTC AE4.03,as well as the recovery time of neutropenia
The recovery time of neutropenia | six weeks
  Comparison of the recovery time between two groups of Polymorphonuclear neutropenia

SECONDARY OUTCOMES:
The incidence of neutropenia associated with Fever (FN) in patients after chemotherapy | six weeks
  Comparison of the incidence of fever with neutropenia in two chemotherapy cycles between two groups.
The incidence of Peripheral blood thrombocytopenia disease | six weeks
  Comparison of the incidence and duration of thrombocytopenia in two chemotherapy cycles between the two groups according to CTC AE4.03.
The duration of Peripheral blood thrombocytopenia disease | six weeks
  Comparison of the incidence and duration of thrombocytopenia in two chemotherapy cycles between the two groups according to CTC AE4.03.
THE incidence and duration of hemoglobin reduction in peripheral blood | six weeks
  Comparison of the incidence and duration of haemoglobin reduction in two chemotherapy cycles between two groups according to CTC AE4.03.
THE duration of hemoglobin reduction in peripheral blood | six weeks
  Comparison of the incidence and duration of haemoglobin reduction in two chemotherapy cycles between two groups according to CTC AE4.03.
THE incidence and duration of peripheral blood leukocyte reduction | six weeks
  Comparison of the incidence and duration of leukopenia in two chemotherapy cycles between the two groups according to CTC AE4.03.
The duration of peripheral blood leukocyte reduction | six weeks
  Comparison of the incidence and duration of leukopenia in two chemotherapy cycles between the two groups according to CTC AE4.03.
The time when the neutrophils were reduced to the lowest point after chemotherapy | six weeks
  Comparison of the time when the neutrophils were reduced to the lowest point after chemotherapy in two chemotherapy cycles between the two groups.
Neutrophil value of neutrophils in patients with low to lowest level after chemotherapy | six weeks
  Comparison of neutrophil values between two groups when neutrophils were reduced to the lowest point after chemotherapy
MDASI-TCM | six weeks
  Comparison of the TCM syndrome score changes between two groups before and after treatment.(if you want see the scale information ,you can reference to the link:https://www.mdanderson.org/content/dam/mdanderson/documents/Departments-and-Divisions/Symptom-Research/MDASI-TCM_SAMPLE.pdf)
Cancer-related fatigue | six weeks
  Comparison of the degree of fatigue changes between two groups before and after treatment.
rhG-CSF dosage | six weeks
  Comparison of the rhG-CSF dosage between two groups before and after treatment.
Immune Index (optional) | six weeks
  Observed indicators include IL-2, INF, NK cells, CD4 +, CD8 +, divided according to the results increased(After treatment than before treatment to improve ≥ 10%, or returned to normal by the abnormalities), decreased(After treatment than before treatment decreased ≥ 10%, or from normal to abnormal changes), stable(After treatment than before treatment, decreased less than 10% or maintained within the normal range).

OTHER OUTCOMES:
Genetic Testing | six weeks
  The changes of body index before and after treatment were compared between two groups of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Hongsheng Lin, Professor, Principal Investigator — CHINA ACADENY OF CHINESE MEDICAL SCIENCES Guang'anmen Hospital
Locations (1):
- CHINA ACADENY OF CHINESE MEDICAL SCIENCES Guang'anmen Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- See also: Standards for the diagnosis and treatment of primary lung cancer (2015 version) in China — http://xueshu.baidu.com/s?wd=paperuri%3A%288f20f17d60dfadfbf49bfa72eef1dc38%29&filter=sc_long_sign&tn=SE_xueshusource_2kduw22v&sc_vurl=http%3A%2F%2Fdoi.med.wanfangdata.com.cn%2Fqk%2Fzhzl201501014&ie=utf-8&sc_us=1930548602497734534
- See also: NCCN Guidelines® : China Editions — http://www.nccnchina.org/nccn-guidelines-china.aspx